CLINICAL TRIAL: NCT02602769
Title: Whole Transcriptome Profiling and Metabolic Phenotyping in Children With ROHHAD Syndrome
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); ROHHAD Association (Unknown)
Responsible Party: Principal Investigator, Vidhu V. Thaker, Assistant Professor, Columbia University
Other Study IDs: AAAS4650; P00018387 (Other: Boston Children's Hospital); R21DK129893 (NIH)
Record Dates: First submitted 2015-11-07; First posted 2015-11-11 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Childhood Obesity; Morbid Obesity
Keywords: Hypoventilation syndrome; Hypothalamic dysfunction; Autonomic dysregulation; Rapid onsey obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity, Morbid; Hypothalamic Diseases; Primary Dysautonomias | interventions — Transcriptome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will retain blood samples for future measurement of hormones involved in regulation of weight, appetite and satiety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases of ROHHAD syndrome: Children diagnosed with ROHHAD syndrome during the course of their clinical care by their physicians.
  The investigators will perform transcriptome profiling in this group.
  Interventions: Diagnostic Test: Transcriptome profiling
- Control cohort: Unaffected first degree family members. The investigators will perform transcriptome profiling in this group.
  Interventions: Diagnostic Test: Transcriptome profiling

INTERVENTIONS:
Diagnostic Test: Transcriptome profiling — The investigators will obtain blood to extract peripheral mononuclear cells. These cells will be used to generate patient specific hypothalamic cells that will be used for transcriptome profiling.

SUMMARY:
Rapid onset Obesity, Hypoventilation, Hypothalamic dysfunction and Autonomic Dysregulation (ROHHAD) is a syndrome named in 2007. The hallmark of the syndrome is the rapid onset obesity and dysregulation of central ventilation. There is little information about the metabolic changes that lead to the rapid onset obesity in these children. The investigators would like to study the metabolic phenotype of these children to understand the disturbances in energy balance that lead to the rapid onset obesity.

DETAILED DESCRIPTION:
Late-onset hypoventilation syndrome with hypothalamic dysfunction was first described in 1965 and renamed to ROHHAD syndrome in 2007 by Ize-Ludlow et al.

The hallmark of ROHHAD syndrome is rapid-onset obesity starting at approximately 1.5 years of age with weight gain of 12-20 kg/year, central hypoventilation distinct from the obstructive hypoventilation caused by obesity, hyperphagia, a spectrum of pituitary hormonal dysfunction, and autonomic disturbances including temperature, blood pressure, and nociception abnormalities. Some children have been noted with developmental and behavioral abnormalities. Tumors of neural crest origin have been identified in 25-33% of the patients. The etiology of ROHHAD syndrome and the cause of rapid onset obesity is unknown.

The aims of this study are to understand the whole transcriptome profiling of patient specific induced pluripotent cell (iPSC) derived hypothalamic neurons to understand the transcriptional level changes that give rise to the manifestations seen in ROHHAD syndrome.

Aim 1. Generate patient specific iPSC-derived hypothalamic neurons from children with ROHHAD syndrome and their unaffected first degree relatives.

Aim 2: Compare the whole transcriptome profiling of the patient derived cells compared to those of unaffected relatives and reference datasets to understand the differences in transcriptome that gives rise to ROHHAD syndrome.

Aim 3: Selected patients may be invited to participate for detailed metabolic phenotyping to understand the mechanisms of excessive weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Children with ROHHAD syndrome

Exclusion Criteria:

* Children with known genetic causes of obesity

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with ROHHAD (Rapid onset Obesity, Hypoventilation, Hypothalamic dysfunction, Autonomic Disturbances), and their first degree relatives.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the transcriptome profile of hypothalamic cells of children with ROHHAD syndrome compared to their unaffected first degree relatives. | 2 year
  The investigators will perform whole transcriptome profiling of iPSC-derived hypothalamic neurons and compare the whole genome sequencing to identify the changes that may give rise to the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Vidhu Thaker, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, New York
  - Columbia University Irving Medical Center, New York, New York

REFERENCES:
- [Result] Thaker VV, Esteves KM, Towne MC, Brownstein CA, James PM, Crowley L, Hirschhorn JN, Elsea SH, Beggs AH, Picker J, Agrawal PB. Whole exome sequencing identifies RAI1 mutation in a morbidly obese child diagnosed with ROHHAD syndrome. J Clin Endocrinol Metab. 2015 May;100(5):1723-30. doi: 10.1210/jc.2014-4215. Epub 2015 Mar 17. PMID 25781356